CLINICAL TRIAL: NCT06198036
Title: Comparative Effects of Hold-Relax and Muscle Energy Techniques for Hamstring Flexibility In School Going Children
Brief Title: Effects of Hold-Relax and Muscle Energy Techniques for Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0733
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Child Development
Keywords: METs; Hamstring flexibility; School going children

STUDY DESIGN:
Intervention Model Description: The study will be Randomized Clinical Trial to compare between the immediate effects of hold-relax Proprioceptive Neuromuscular Facilitation and Muscle Energy Technique (RI) for hamstring flexibility in school. Participants meeting the pre-determind inclusion and exclusion criteria will be divided into two groups going children
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Application of Hold-Relax PNF Technique (Active Comparator): A hold-relax technique that entails stretching the muscle to its maximum length. Participant will be in supine position. The hamstring muscle will be stretched for 7 to 10 seconds while the individual reported only a slight stretch in the muscle. The participant then attempts to lower his leg towards the table while being resisted by the researcher, isometrically contracting his hamstring muscle for 3 seconds. The patient then instructed to relax for five seconds. The researcher then passively stretched the muscle until a slight sensation of stretch was experienced. The stretch will maintain for seven seconds. There were five repetitions of this sequence, each one 20 seconds apart from the previous one
  Interventions: Other: Hold-Relax Technique
- Group B: Application of Muscle Energy Technique (Active Comparator): Group B will receive a Muscle Energy Technique (MET) applying the reciprocal inhibition principle. Participant will be in supine lying and the affected muscle held in a mid-range position. The Reciprocal Inhibition-MET group stretched for 10 to 60 seconds after performing an isometric contraction of the muscle opposite the one that needed to be stretched for 7 to 10 seconds (30%-50% of the time) followed by 5 second rest interval. With a pause of 20 seconds in between each repetition, this sequence was performed five times(52). The readings for Active knee Extension (AKE), TUG test and WBFPS before and after treatment session determined the improvement regarding the treatment outcomes.
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Hold-Relax Technique — Participants in this group will be treated with hold-relax PNF Technique
  Arms: Group A: Application of Hold-Relax PNF Technique
Other: Muscle Energy Technique — Participants in this group will be treated with Muscle Energy Technique via Reciprocal Inhibition Mechanism
  Arms: Group B: Application of Muscle Energy Technique

SUMMARY:
The most important aspect of physical fitness is flexibility, which can be greatly impacted by bad posture. Long periods of sitting in school going children can cause the hamstring muscles to shorten because they bend the knee. There are numerous methods for improving hamstring flexibility, but very few of them produce immediate results. The purpose of this study will be to compare between the immediate effects of hold-relax proprioceptive neuromuscular facilitation and muscle energy technique (MET) for hamstring flexibility in school going children. This will be the randomized clinical trial in which total time of six month will be utilized after the approval from BASR. Data will be collected from Unique Science School Al-Rehman Campus, Lahore. 106 participants will be taken with 05-12 years of age through purposive sampling technique. Participants will be divided into two equal groups. Participants in group A will be given hold-relax PNF and the group B will underwent METs (reciprocal inhibition). Hamstring ROM will be assessed through AKET. Measurements will be taken by goniometer. Wong-Baker faces pain scale (WBFPS) and Timed 'Up and Go' (TUG) test will be used to evaluate pain and functional mobility respectively. Data will be analyzed on SPSS version 25. Results after statistical analysis will show which technique is more effective and will have best outcomes.

DETAILED DESCRIPTION:
The most important aspect of physical fitness is flexibility, which can be greatly impacted by bad posture that might occur from a sedentary lifestyle of a person and a reduction in the soft tissues' flexibility cause serious musculoskeletal injuries. Long periods of sitting in school going children can cause the hamstring muscles to shorten because they bend the knee. There are numerous methods for improving hamstring flexibility, but very few of them produce immediate results. The literature demonstrated that the two most successful stretching methods to compare were hold-relax and MET but there is paucity to determine their immediate effectiveness.

The purpose of this study will be to compare between the immediate effects of hold-relax proprioceptive neuromuscular facilitation and muscle energy technique (MET) for hamstring flexibility in school going children and to determine which strategy improves hamstring flexibility in school-aged children the fastest and with the best results. This will be the randomized clinical trial in which total time of six month will be utilized after the approval from BASR. Data will be collected from Unique Science School Al-Rehman Campus, Lahore. 106 participants will be taken with 05-12 years of age through purposive sampling technique. Participants will be divided into two equal groups. Participants in group A will be given hold-relax PNF and the group B will underwent METs (reciprocal inhibition). Hamstring ROM will be assessed through AKET. Measurements will be taken by goniometer. Wong-Baker faces pain scale (WBFPS) and Timed 'Up and Go' (TUG) test will be used to evaluate pain and functional mobility respectively. Data will be analyzed on SPSS version 25. Results after statistical analysis will show which technique is more effective and will have best outcomes

ELIGIBILITY:
Inclusion Criteria

* Age 5-12 years children
* Gender (both male and female)
* Normal children
* Hamstring tightness (minimum degree <160 degrees

Exclusion Criteria

* Regular athletes
* Past pathology
* Post fracture of limb
* Leg length discrepancy
* History of spinal cord injury
* Presence of physical deformities
* Subject not willing to participate
* Subject using lower limb prosthesis or orthotic device

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Goniometer | eight weeks
  The universal full circle goniometer is arguably the preferred instrument for measuring ROM for the majority of applications to the extremities. This version, which has a body, moving arm, and stationary arm, is the most prevalent. When comparing radiographic measurements with goniometric measurements in sedated and unsedated cats, joint measurements did not change significantly by measurement type. Cronbach alpha values for goniometric joint measurements were more than 0.99.
Active Knee Extension Test (AKET) | eight weeks
  The Active Knee Extension Test measures the range of active knee extension when the hip is flexed as well as the length of the hamstring muscles. If the body positions are sufficiently stable, this test has a high degree of reliability. This test, a self-monitored variation of the active knee extension test, has also proven to be successful when performed by the person being tested. Among healthy individuals, the inter-rater and intra rater dependability has been proven.

SECONDARY OUTCOMES:
Wong Baker Faces Pain Scale (WBFPS) | Eight weeks
  The Wong Baker Faces Pain Scale is a self-report tool designed to determine how much pain children are experiencing. Using scales of various facial expressions and matching a child's pain level to a similar face is one method of measuring pain in children. The Faces scale is an ordinal outcome measure that contains a minimal and predetermined number of categorical responses that are presented in a predetermined pattern. It is used to measure the rating of pain.
Timed 'Up and Go' Test (TUG) | Eight Weeks
  The Timed Up and Go test (TUG test), also used to measure functional mobility in children, is a useful tool. The TUG test calculates how long it takes to stand up, go forward 10 feet, turn around, move backward, and then sit down. The TUG test shows strong consistency and correlation with other evaluation instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Sunnia Mudabber, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funk D, Swank AM, Adams KJ, Treolo D. Efficacy of moist heat pack application over static stretching on hamstring flexibility. J Strength Cond Res. 2001 Feb;15(1):123-6. PMID 11708695